CLINICAL TRIAL: NCT01963104
Title: Community-Based Kiosks for Hearing Screening and Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Portland VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, M. Patrick Feeney, Director of NCRAR, Portland VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 4R33DC011769-02 (NIH)
Record Dates: First submitted 2013-09-12; First posted 2013-10-16 (Estimated); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Hearing Loss
Keywords: hearing test, audiology, healthcare utilization,; patient education, hearing screening
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- Automated hearing test (Experimental): Subjects will take an abbreviated automated hearing test and then receive recommendations for hearing healthcare follow-up.
  Interventions: Procedure: Automated hearing test
- Pure-tone Screener test (Experimental): Subjects will take a pure-tone hearing screening test and then receive recommendations for hearing healthcare follow-up.
  Interventions: Procedure: Pure-tone Screener test
- Digits-in-noise test (Experimental): Subjects will take a digits-in-noise test and then receive recommendations for hearing healthcare follow-up.
  Interventions: Procedure: Digits-in-noise test
- No screening test (Experimental): This group of subjects will not receive a screening test.
  Interventions: Procedure: No screening test
- Automated hearing test/Motivation video (Experimental): Subjects will take an abbreviated automated hearing test and then receive recommendations for hearing healthcare follow-up. They will then watch a brief video that shows how hearing works and learn about the different types of hearing loss.
  Interventions: Procedure: Automated hearing test/Motivation video
- Pure-tone Screener/Motivation video (Experimental): Subjects will take a pure-tone hearing screening test and then receive recommendations for hearing healthcare follow- up. They will then watch a brief video that shows how hearing works and learn about the different types of hearing loss.
  Interventions: Procedure: Pure-tone Screener/Motivation video
- Digits-in-noise test/Motivational video (Experimental): Subjects will take a digits-in-noise test and then receive recommendations for hearing healthcare follow-up.They will then watch a brief video that shows how hearing works and learn about the different types of hearing loss.
  Interventions: Procedure: Digits-in-noise test/Motivational video
- No screening test/Motivational video (Experimental): This group of subjects will not receive a screening test. They will watch a brief video that shows how hearing works and learn about the different types of hearing loss
  Interventions: Procedure: No screening test/Motivational video
- Home Hearing Screening Test (Experimental): Subjects will be taught the set-up for a home hearing screening test, take an abbreviated automated hearing test and then receive recommendations for hearing healthcare follow-up.
  Interventions: Procedure: Home Hearing Screening Test
- Home Hearing Screening Test/Brief video (Experimental): Subjects will be taught the set-up for a home hearing screening test, take an abbreviated automated hearing test and then receive recommendations for hearing healthcare follow-up.
  They will then watch a brief video that shows how hearing works and learn about the different types of hearing loss.
  Interventions: Procedure: Home Hearing Screening Test/Brief video

INTERVENTIONS:
Procedure: Automated hearing test — Subjects will take an automated hearing test that presents tones at different pitches and volumes. Participants will identify whether or not they heard the tone and receive printed recommendations for hearing healthcare follow-up. All subjects will complete the Hearing Handicap Inventory (HHI) questionnaire and the Hearing Beliefs Questionnaire (HBQ). Approximately 6-8 months after their initial appointment, subjects in this groups will receive a telephone call and will be asked questions related to their actions and attitudes related to hearing and hearing health care.
  Arms: Automated hearing test
Procedure: Pure-tone Screener test — During the test different tones are going to be presented at one volume level. Participants will identify whether or not they heard the tone and receive printed recommendations for hearing healthcare follow-up. All subjects will complete the Hearing Handicap Inventory (HHI) questionnaire and the Hearing Beliefs Questionnaire (HBQ). Approximately 6-8 months after their initial appointment, subjects in this groups will receive a telephone call and will be asked questions related to their actions and attitudes related to hearing and hearing health care.
  Arms: Pure-tone Screener test
Procedure: Digits-in-noise test — During the test subjects will hear a pattern of 3 numbers with variable noise in the background and identify the pattern they hear, and receive printed recommendations for hearing healthcare follow-up. All subjects will complete the Hearing Handicap Inventory (HHI) questionnaire and the Hearing Beliefs Questionnaire (HBQ). Approximately 6-8 months after their initial appointment, subjects in this groups will receive a telephone call and will be asked questions related to their actions and attitudes related to hearing and hearing health care.
  Arms: Digits-in-noise test
Procedure: No screening test — This group of subjects will not receive a screening test. All subjects will complete the Hearing Handicap Inventory (HHI) questionnaire and the Hearing Beliefs Questionnaire (HBQ). Approximately 6-8 months after their initial appointment, subjects in this group will receive a telephone call and will be asked questions related to their actions and attitudes related to hearing and hearing health care.
  Arms: No screening test
Procedure: Automated hearing test/Motivation video — Subjects will take an automated hearing test that presents tones at different pitches and volumes.Participants will identify whether or not they heard the tone and receive printed recommendations for hearing healthcare follow-up. They will also watch a brief video that shows how hearing works and learn about the different types of hearing loss. All subjects will complete the Hearing Handicap Inventory (HHI) questionnaire and the Hearing Beliefs Questionnaire (HBQ). Approximately 6-8 months after their initial appointment, subjects in this groups will receive a telephone call and will be asked questions related to their actions and attitudes related to hearing and hearing health care.
  Arms: Automated hearing test/Motivation video
Procedure: Pure-tone Screener/Motivation video — During the test different tones are going to be presented at one volume level. Participants will identify whether or not they heard the tone and receive printed recommendations for hearing healthcare follow-up. They will also watch a brief video that shows how hearing works and learn about the different types of hearing loss. All subjects will complete the Hearing Handicap Inventory (HHI) questionnaire and the Hearing Beliefs Questionnaire (HBQ). Approximately 6-8 months after their initial appointment, subjects in this group will receive a telephone call and will be asked questions related to their actions and attitudes related to hearing and hearing health care.
  Arms: Pure-tone Screener/Motivation video
Procedure: Digits-in-noise test/Motivational video — During the test subjects will hear a pattern of 3 numbers with variable noise in the background and identify the pattern they hear, and receive printed recommendations for hearing healthcare follow-up. They will also watch a brief video that shows how hearing works and learn about the different types of hearing loss. All subjects will complete the Hearing Handicap Inventory (HHI) questionnaire and the Hearing Beliefs Questionnaire (HBQ). Approximately 6-8 months after their initial appointment, subjects in this group will receive a telephone call and will be asked questions related to their actions and attitudes related to hearing and hearing health care.
  Arms: Digits-in-noise test/Motivational video
Procedure: No screening test/Motivational video — This group of subjects will not receive a screening test. They will watch a brief video that shows how hearing works and learn about the different types of hearing loss. All subjects will complete the Hearing Handicap Inventory (HHI) questionnaire and the Hearing Beliefs Questionnaire (HBQ). Approximately 6-8 months after their initial appointment, subjects in this group will receive a telephone call and will be asked questions related to their actions and attitudes related to hearing and hearing health care.
  Arms: No screening test/Motivational video
Procedure: Home Hearing Screening Test — Subjects will be taught the set-up for a home hearing screening test and will take an automated hearing test that presents tones at different pitches and volumes. Participants will identify whether or not they heard the tone and receive printed recommendations for hearing healthcare follow-up. All subjects will complete the Hearing Handicap Inventory (HHI) questionnaire and the Hearing Beliefs Questionnaire (HBQ). Approximately 6-8 months after their initial appointment, subjects in this groups will receive a telephone call and will be asked questions related to their actions and attitudes related to hearing and hearing health care.
  Arms: Home Hearing Screening Test
Procedure: Home Hearing Screening Test/Brief video — Subjects will be taught the set-up for a home hearing screening test and will take an automated hearing test that presents tones at different pitches and volumes. Participants will identify whether or not they heard the tone and receive printed recommendations for hearing healthcare follow-up. All subjects will complete the Hearing Handicap Inventory (HHI) questionnaire and the Hearing Beliefs Questionnaire (HBQ). They will also watch a brief video that shows how hearing works and learn about the different types of hearing loss.
  Approximately 6-8 months after their initial appointment, subjects in this groups will receive a telephone call and will be asked questions related to their actions and attitudes related to hearing and hearing health care.
  Arms: Home Hearing Screening Test/Brief video

SUMMARY:
The overall goal of the project is to evaluate innovative, cost-effective, community-based automated hearing screening and education methods to motivate individuals with mild-to-moderate hearing loss to enter the hearing healthcare system.

ELIGIBILITY:
Inclusion Criteria: :

* Some subjects will have a complaint of hearing difficulty without a recent hearing evaluation

Exclusion Criteria:

* For all groups: minimum age 18 years. No current hearing aid use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2048 (Actual)
Dates: Start 2013-09; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Record number of participants who sought hearing healthcare 6 months after the initial visit. | 4 years

SECONDARY OUTCOMES:
Record number of participants whose attitude about hearing health care has changed 6 months after the initial visit. | 4 years

OTHER OUTCOMES:
Record which hearing screening method was best at motivating subjects to pursue hearing healthcare. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Martin P Feeney, Ph.D., Principal Investigator — Portland VA Medical Center, National Center for Rehabilitative Auditory Research
Locations (4):
- United States (4):
  - Bay Pines VAHCS, Bay Pines, Florida
  - University of Minnesota, Minneapolis, Minnesota
  - Ohio State University, Columbus, Ohio
  - Portland VA Medical Center, National Center for Rehabilitative Auditory Research, Portland, Oregon